CLINICAL TRIAL: NCT07133971
Title: A Clinical Observational Study Evaluating the Efficacy of Cerave Neuroceramide Intensive Repair Body Lotion in Improving Dry Skin in the Elderly
Brief Title: A Clinical Observational Study Evaluating the Efficacy of Cerave Neuroceramide Intensive Repair Body Lotion .
Status: Not yet recruiting | Type: Observational
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Other Study IDs: C25005056
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Dry Skin in the Elderly

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with moderate to severe skin dryness: Based on ODS and NRS scores, patients with moderate to severe skin dryness (moderate-grade 2, severe-grade 3) were assessed.
  Interventions: Other: skin care product（Cerave Neuroceramide Moisturizing Repair Body Lotion）

INTERVENTIONS:
Other: skin care product（Cerave Neuroceramide Moisturizing Repair Body Lotion） — All study participants will use Cerave Neuroceramide Moisturizing Body Lotion during the trial period, applying it every night to dry skin areas. If topical medications are used, they should be applied first to dry skin areas, followed by the product.

SUMMARY:
This study is a single-center observational clinical study aimed at evaluating the impact of Cerave Neuroceramide Moisturizing Repair Body Lotion on the quality of life, improvement in skin condition, and satisfaction with the product experience among individuals with moderate to severe dry skin associated with aging. The study plans to recruit approximately 210 male or female participants aged 55 years or older with moderate to severe skin dryness in the affected areas (accounting for a dropout rate and protocol violation rate of no more than 5%), and will screen participants based on inclusion and exclusion criteria to ensure that at least 200 participants complete the study. Participants entering this study will be categorized based on ODS and NRS scores into: moderate or severe skin dryness (moderate-grade 2, severe-grade 3), with the sample size ratio between moderate and severe groups maintained at 1:1. This study will last for 4 weeks and include 2 visits. Visits will be conducted at baseline (T0) and week 4 (T4w). The window period for the week 4 (T4w) visit is ±2 days. This study does not involve randomization. All study participants will use Cerave Neuroceramide Moisturizing Repair Body Lotion on areas of skin dryness.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with moderate to severe skin dryness as assessed by a clinician (ODS score of 2 or 3)
* Individuals with moderate to severe self-reported skin itching as assessed by a clinician (NRS ≥ 1)
* Individuals aged 55 years and older
* Open to patients with one or more of the following conditions:

  1. History of atopic dermatitis;
  2. Currently using a stable medication regimen prescribed and monitored by a physician (ongoing use), where the medication has side effects causing skin dryness (e.g., statins, calcium channel blockers, diuretics, antiplatelet agents, ACE inhibitors, beta-blockers, adrenergic receptor agonists, immunosuppressants, etc.);
  3. Patients with systemic diseases associated with dryness (diagnosed and managed by a physician), such as diabetes, hyperthyroidism, hypothyroidism, or hemodialysis.
* Voluntarily participate in the trial, understand and agree to sign the informed consent form, and agree to follow the study protocol throughout the study period, including using the study-provided products, not using other similar products, completing a diary, and attending regular follow-up visits as required by the trial.

Exclusion Criteria:

* Individuals with a history of allergy, allergic reaction, or hypersensitivity to any component of the study product (Cerave Neuroceramide Moisturizing Repair Body Lotion);
* Individuals with a history of allergic contact dermatitis secondary to the use of moisturizing products;
* Individuals with any clinical manifestations or other conditions at the treatment site that the physician deems may affect the evaluation or results of the study product;
* Individuals who are unable or unwilling to attend all study visits and adhere to the treatment regimen;
* Individuals who have participated in any other drug clinical studies within the past 3 months prior to the start of the trial.

Min Age: 55 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male or female study participants aged 55 years or older with moderate to severe skin dryness.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-08-22 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Changes in ODS grading before and after using the trial product | Baseline visit, Week 4 visit
  The Overall Dry Skin Score (ODS) is used to comprehensively assess the severity of objective findings of skin dryness. The following are the skin manifestations and scores for ODS grading:
  A score of 0 indicates no dryness symptoms, smooth skin, no scaling, no roughness, no erythema, and no fissures； Score 1 indicates mild dryness, occasional scaling, uneven distribution, and slightly rough and dull skin appearance； Score 2 indicates moderate dryness, with small flakes or small patches of scales on the skin surface, and mildly rough and whitish appearance； Score 3 indicates severe dryness, with evenly distributed scales, a noticeably rough skin appearance, mild redness, and minor cracks； Score 4 indicates extremely severe dryness, with extensive scale shedding, a rough and reddened skin appearance accompanied by eczema-like changes and fissures.
Changes in NRS scores before and after use of the trial product | Baseline visit, Week 4 visit
  The NRS itch score ranges from 0 (no itching) to 10 (severe itching). Clinicians ask participants to verbally express the severity of their subjective itching using numerical values. The following are reference values for the NRS itch score:
  Score 0 indicates no itching Score 1-2 indicates mild itching Score 3-6 indicates moderate itching Score 7-8 indicates severe itching Score 9-10 indicates very severe itching
Doctors assess the skin condition of participants by completing a scoring form | Baseline visit, week 4 visit
  Doctors assess the skin condition of participants by completing a scoring form, which uses a 0-4 point scale (0 points indicating no symptoms, 4 points indicating severe symptoms). The form includes the following criteria: skin dryness, skin flaking/peeling/scaling, skin roughness, skin redness/erythema, skin cracking, and noticeable irritation caused by scratching.
Quality of life self-assessment questionnaire completed by subjects | Baseline visit, Week 4 visit
  Subjects completed a quality of life self-assessment questionnaire using a 1-4 point scale (1 point indicating none at all, 4 points indicating to a great extent), which included questions on whether subjects felt depressed, embarrassed, or stressed due to dry skin, and whether dry skin affected subjects' daily lives, social activities, etc.

SECONDARY OUTCOMES:
Doctors assess participants' tolerance and satisfaction with the trial product by completing a questionnaire | Week 4 visit
  Doctors assess the trial product's tolerance by completing a questionnaire, which is a 1-4 point rating scale (1 = low, 4 = very high). Doctors assess overall satisfaction with the trial product by completing a questionnaire, which is a 1-5 point rating scale (1 = very dissatisfied, 5 = very satisfied).
Patient self-assessment questionnaire for tolerability and satisfaction with the investigational product | Week 4 visit
  Patients assess the tolerability of the trial product by completing a questionnaire, which is a 1-4 point rating scale (1 = low, 4 = very high). Patients assess their overall satisfaction with the trial product by completing a questionnaire, which is a 1-5 point rating scale (1 = very dissatisfied, 5 = very satisfied).
Cosmetic characteristics questionnaire completed by patients | Week 4 vist
  Patients complete a cosmetic characteristics questionnaire, which mainly includes questions about absorption, stickiness, smell, texture, feel, and whether it makes the skin feel comfortable. The questionnaire is scored on a scale of 1 to 5, with 1 = completely disagree and 5 = completely agree.